CLINICAL TRIAL: NCT03716180
Title: DAPHNe: De-escalation to Adjuvant Antibodies Post-pCR to Neoadjuvant THP (Paclitaxel/Trastuzumab/Pertuzumab)-a Pilot Study in HER2-positive Breast Cancer
Brief Title: DAPHNe: Paclitaxel/Trastuzumab/Pertuzumab in HER2-Positive BC
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Susan G. Komen Breast Cancer Foundation (Other); Breast Cancer Research Foundation (Other); Terri Brodeur Breast Cancer Foundation (Unknown)
Responsible Party: Principal Investigator, Adrienne G. Waks, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-394
Record Dates: First submitted 2018-10-19; First posted 2018-10-23 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer
Keywords: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Paclitaxel; Trastuzumab; pertuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Paclitaxel+Trastuzumab+Pertuzumab (Experimental): Paclitaxel is administered intravenously on days 1, 8, and 15 of each 21-day cycle Trastuzumab is administered intravenously on day 1 of each 21-day cycle Pertuzumab is administered intravenously on Day 1 of each 21-day cycle
  Interventions: Drug: Paclitaxel; Drug: Trastuzumab; Drug: Pertuzumab

INTERVENTIONS:
Drug: Paclitaxel — Paclitaxel is an anti-cancer ("antineoplastic" or "cytotoxic") chemotherapy drug
  Other Names: Taxol
Drug: Trastuzumab — Trastuzumab works by targeting the HER2/neu receptor on cancer cells
  Other Names: Herceptin
Drug: Pertuzumab — Pertuzumab is a monoclonal antibody which targets the surface of the cells human epidermal growth factor receptor 2 protein (HER2) on the cancer cell, interfering with HER2 causing cancer cell death
  Other Names: Perjeta

SUMMARY:
This research study is studying whether participants and their doctors are willing to determine post-surgery treatment on the basis of response to pre-surgery treatment, and studying blood and tissue collected from participants treated with a combination of drugs as a treatment for breast cancer.

The names study drugs involved in this study are:

* Paclitaxel (also called Taxol)
* Trastuzumab (also called Herceptin)
* Pertuzumab (also called Perjeta)

DETAILED DESCRIPTION:
This research study is a Pilot Study, which means investigators are looking at the feasibility of a new approach for deciding the optimal medical treatment for this type of breast cancer. The FDA (the U.S. Food and Drug Administration) has approved paclitaxel, trastuzumab, and pertuzumab as part of a pre-operative treatment option for this disease.

The purpose of this study is to evaluate whether participants and their doctors are willing to accept a treatment recommendation for post-operative chemotherapy, on the basis of the participant's response to pre-operative treatment with paclitaxel, trastuzumab, and pertuzumab.

In addition, the investigators are evaluating how the body's immune system works with paclitaxel, trastuzumab, and pertuzumab to kill cancer cells. For this reason, the investigators will collect samples of the participant's breast tumor and samples of the participant's blood over time to understand the reaction of the immune system to the participant's tumor.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have Stage II or III (according to AJCC cancer staging manual anatomic staging table, 8th edition) histologically confirmed invasive carcinoma of the breast. A minimum tumor size of 1.5 cm determined by physical exam or imaging (whichever is larger) is required. Patients with inflammatory breast carcinoma (T4d) are NOT eligible.
* Tumors must be HER-2 positive, as assessed by standard local institutional protocol (central testing is not required):

  * IHC 3+
  * FISH positive based on one of the three following criteria:

Single-probe average HER2 copy number ≥ 6.0 signals/cell; OR

* Dual-probe HER2/CEP17 ratio <2.0 with an average HER2 copy number ≥ 6.0 signals/cell; OR
* Dual-probe HER2/CEP17 ratio ≥2.0

  * ER/PR determination is required. ER- and PR-assays should be performed by immunohistochemical methods according to the local institution standard protocol.
  * Bilateral breast cancers are allowed as long as both cancers are HER2-positive (as defined in 3.1.2), or the contralateral cancer is a <1 cm, ER+, and HER2- tumor.
  * Patients with multifocal or multicentric disease are eligible as long as all tumor foci that were tested for HER2 status at the local institution are HER2-positive, and at least one tumor focus meets eligibility criteria.
  * Breast imaging should include dedicated ultrasound of the ipsilateral axilla. For subjects with a clinically positive axilla based on exam or imaging, a fine needle aspiration or core biopsy procedure will be performed to determine the presence of metastatic disease in the lymph nodes (though lymph node sampling procedure need not be resulted prior to patient's registration on trial, as long as all other eligibility are met).
  * Men and women (with any menopausal status) ≥ 18 years of age are eligible.
  * ECOG PS 0 or 1.
* Required laboratory values:
* ANC ≥ 1000/mm3
* Hemoglobin ≥ 9 g/dl
* Platelets ≥ 100,000/mm3
* Serum creatinine < 1.5 x ULN (institutional) OR calculated GFR ≥60mL/min.

  -Total bilirubin ≤ 1.5 x ULN (institutional). For patients with Gilbert Syndrome, the direct bilirubin should be within the institutional normal range OR total bilirubin ≤ 2.0 mg/dL.
* AST and ALT ≤ 2.5x ULN (institutional)

  * Left ventricular ejection fraction (LVEF) ≥ 50%.
  * Premenopausal women must have a negative serum pregnancy test within 14 days of registration, including women who have had a tubal ligation and for women less than 12 months after the onset of menopause.
  * Women of childbearing potential and men with partners of childbearing potential must be willing to use one highly effective form of non-hormonal contraception or two effective forms of non-hormonal contraception by the patient and/or partner and continue its use for the duration of the study treatment and for 7 months after the last dose of study treatment.
  * Patients with a history of ipsilateral DCIS are eligible.
  * Patients undergoing breast conservation therapy (i.e. lumpectomy) must not have any contraindications to radiation therapy.
  * Willing and able to sign informed consent.
  * Willing to provide tissue for research purposes

Exclusion Criteria:

* Pregnant or nursing women due to the teratogenic potential of the study drugs.
* Active, unresolved infection.
* Receipt of intravenous antibiotics for infection within 7 days prior to registration.
* Uncontrolled hypertension (systolic >180 mm Hg and/or diastolic >100 mm Hg) or clinically significant (i.e. active) cardiovascular disease: cerebrovascular accident/stroke or myocardial infarction within 6 months prior to first study medication, unstable angina, congestive heart failure (CHF) of New York Heart Association (NYHA) Class II or higher (see Appendix B), or serious cardiac arrhythmia requiring medication.
* Significant symptoms (Grade ≥ 2) from peripheral neuropathy.
* Other concurrent serious diseases that may interfere with planned treatment, including severe pulmonary conditions/illness, uncontrolled infections, uncontrolled diabetes.
* Any prior treatment for the current breast cancer, including chemotherapy, hormonal therapy, radiation, or experimental therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-11-05 (Actual); Primary Completion 2020-10-08 (Actual); Study Completion 2030-09-01 (Estimated)

PRIMARY OUTCOMES:
Adjuvant chemotherapy Received | 2.5 years
  To assess adherence to protocol-specified antibody doublet therapy in the adjuvant setting among patients with stage II-III HER2+ breast cancer who achieve pathologic complete response (pCR) following neoadjuvant Paclitaxel/Trastuzumab/Pertuzumab (THP).

SECONDARY OUTCOMES:
pCR rate | 2 years
  To assess pathologic complete response (pCR) for 1) all patients, 2) hormone receptor positive (HR+) patients, and 3) hormone receptor negative (HR-) patients
Residual Cancer Burden (RCB) scores | 2 years
  To assess residual cancer burden (RCB) in 1) all patients, 2) hormone receptor positive patients (HR+), 3) hormone receptor negative (HR-) patients. RCB is scored from 0 to 3, (with possible values 0, 1, 2, 3), where 0 is the best score and indicates eradication of all disease at the time of surgery, and 3 is the worst score, indicating poor response to preoperative therapy.
Reasons for Off-Protocol Escalation per study-specific questionnaires | 2 years
  Patients and physicians will complete questionnaires to assess reasons for off-protocol escalation (meaning, a decision to administer post-operative chemotherapy, for patients with pCR). Standardized questionnaires for both patients and physician reviewers have been developed specifically for this study. Responses are qualitative and do not involve a scale.
Reasons for Off-Protocol De-Escalation per study-specific questionnaires | 2 years
  Patients and physicians will complete questionnaires to assess reasons for off-protocol de-escalation (meaning, a decision not to administer post-operative chemotherapy, for patients without pCR). Standardized questionnaires for both patients and physician reviewers have been developed specifically for this study. Responses are qualitative and do not involve a scale.
One Year of Trastuzumab and Pertuzumab | 3 years
  To assess the percentage of patients completing one year of HP
Event-Free Survival (EFS) | 12 years
  To measure event-free survival (EFS), and to compare EFS in the following subgroups: 1) Patients with pCR versus patients without pCR; 2) Patients with RCB 0 or 1, versus patients with RCB 2 or 3
Recurrence-Free Interval (RFI) | 12 years
  To measure recurrence-free interval (RFI), and to compare RFI in the following subgroups: 1) Patients with pCR versus patients without pCR; 2) Patients with RCB 0 or 1, versus patients with RCB 2 or 3
Overall survival (OS) | 12 years
  To measure overall survival (OS) as an exploratory endpoint
Post-THP (Paclitaxel/Trastuzumab/Pertuzumab) imaging findings and pathology findings in the surgical specimen | 2 years
  To evaluate correlation between post-THP (Paclitaxel/Trastuzumab/Pertuzumab) imaging findings and pathology findings in the surgical specimen

CONTACTS AND LOCATIONS:
Overall Officials: Adrienne G Waks, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (5):
- United States (5):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - DF/BWCC at Milford Regional Medical Center, Milford, Massachusetts
  - DF/BWCC in clinical affiliation with South Shore Hospital, South Weymouth, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Weiss A, Li T, Desai NV, Tung NM, Poorvu PD, Partridge AH, Nakhlis F, Dominici L, Sinclair N, Spring LM, Faggen M, Constantine M, Krop IE, DeMeo M, Wrabel E, Alberti J, Chikarmane S, Tayob N, King TA, Tolaney SM, Winer EP, Mittendorf EA, Waks AG. Impact of Neoadjuvant Paclitaxel/Trastuzumab/Pertuzumab on Breast Tumor Downsizing for Patients with HER2+ Breast Cancer: Single-Arm Prospective Clinical Trial. J Am Coll Surg. 2023 Aug 1;237(2):247-256. doi: 10.1097/XCS.0000000000000761. Epub 2023 May 17. PMID 37194964
- [Derived] Waks AG, Desai NV, Li T, Poorvu PD, Partridge AH, Sinclair N, Spring LM, Faggen M, Constantine M, Metzger O, Alberti J, Deane J, Rosenberg SM, Frank E, Tolaney SM, Krop IE, Tung NM, Tayob N, King TA, Mittendorf EA, Winer EP. A prospective trial of treatment de-escalation following neoadjuvant paclitaxel/trastuzumab/pertuzumab in HER2-positive breast cancer. NPJ Breast Cancer. 2022 May 10;8(1):63. doi: 10.1038/s41523-022-00429-7. PMID 35538105